CLINICAL TRIAL: NCT06326606
Title: A Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MLS101 (psilocybin) in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of MLS101 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MycoMedica Life Sciences PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-MLS101-101
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, single ascending and multiple dose study to assess the safety, tolerability, and pharmacokinetics of MLS101 in healthy participants.
  Single Ascending Dose (SAD): 24 participants will be enrolled in 3 sequential dose cohorts and will be randomized to receive a single dose of MLS101 or placebo. Additional cohorts (comprising 8 participants in each cohort) may be enrolled to explore more doses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MLS101 (Active Comparator): MLS101 capsule(s) administered orally as a once a day dose
  Interventions: Drug: Psilocybin
- Placebo (Placebo Comparator): Active treatment matching capsules will be administered orally as a once a day dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Psilocybin — Capsule containing active ingredient, psilocybin
  Other Names: MLS101
  Arms: MLS101
Drug: Placebo — Capsule with no active ingredients
  Arms: Placebo

SUMMARY:
MLS101 is being developed as a low dose psilocybin, that can be administered to treat various neurological and psychiatric conditions.

The purpose of this clinical trial is to assess how safe and tolerated MLS101 is; to see how MLS101 is distributed and cleared by the body (pharmacokinetics); and to assess the psychedelic effects of MLS101 in healthy adult participants.

DETAILED DESCRIPTION:
In recent years, high-dose psilocybin has gained attention for its potential therapeutic benefits in many psychiatric indications, however existing clinical data for low psilocybin doses are limited.

Microdoses are generally considered to be those absent of profound sensory and cognitive effects that would interfere with normal everyday functioning, but only a small number of prospective studies have evaluated microdoses and/or low doses in a controlled manner.

As a foundational study of the therapeutic use of low doses of psilocybin, this study will evaluate the safety, tolerability, pharmacokinetics, and sensorial effects using a prospective, controlled, single ascending dose/multiple ascending doses in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females aged 18 to 65 years old (inclusive) at the time of signing the informed consent form. Standard contraception measures are required for this clinical trial.
2. Healthy, in the opinion of the Investigator, based on prior (history of) or current (ongoing) medical and psychiatric screening assessments.
3. Participants with no clinically significant findings on physical examination, laboratory tests, and cardiac assessment.
4. Body mass index (BMI) within the range 18-32 kg/m2, inclusive.
5. Normal blood pressure.
6. Capable of giving signed informed consent which includes the requirements and restrictions as per the approved study protocol.

Key Exclusion Criteria:

1. Prior known exposure to psilocybin within the past 10 years.
2. Prior (history of) or current (ongoing) diagnosis, or first-degree relatives with clinically significant medical or psychiatric condition or disease.
3. History of or presence of cardiovascular disease.
4. Abnormal and clinically significant ECG.
5. History or presence of a neurodegenerative disorder such Alzheimer's disease or Parkinson's disease.
6. Use of medications that have CNS effects or affect performance.
7. Use of medications with serotonergic activity.
8. History or presence of hypersensitivity or idiosyncratic reaction to psilocybin or related compounds.
9. History of substance or alcohol abuse disorder in the last 1 year.
10. Participant who, for any reason, is deemed by the Investigator to be inappropriate for this study; or has any condition which would confound or interfere with the evaluation of the safety, tolerability, or PK of the investigational drug; or is unable to comply with the study protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and seriousness of treatment-emergent adverse events (TEAEs) | Screening (Day -60) to end of study visit (Day 8)
Occurrence of clinically significant changes in physical examination, vital signs, ECGs, clinical laboratory tests, the Columbia-Suicide Severity Rating Scale (C-SSRS). | Screening (Day -60) to end of study visit (Day 8)
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a short questionnaire. If there is a positive result for suicidality on the C-SSRS after Screening (defined by a participant answering "yes" to questions 4 or 5 on the suicidal ideation portion of the C-SSRS), the participant will be evaluated by an Investigator or medically qualified Sub-investigator for continuation in the study. Participants with suicidal ideation or behavior (a "yes" answer at any time during treatment to any one of the ten suicidal ideation and behavior questions (Categories 1-10) on the C-SSRS) at any time during the study will be withdrawn from the study. If a participant becomes suicidal during the study, an Investigator or medically qualified Sub-investigator should provide the appropriate treatment to the participant.

SECONDARY OUTCOMES:
Pharmacokinetics of MLS101: maximum observed serum concentration (Cmax) | Day 1 to Day 3 post-dose and end of study visit (Day 8)
Pharmacokinetics of MLS10: area under the plasma concentration-time curve (AUC) | Day 1 to Day 3 post-dose and end of study visit (Day 8)
Pharmacokinetics of MLS101: time corresponding to the occurrence of Cmax (tmax) | Day 1 to Day 3 post-dose and end of study visit (Day 8)
Pharmacokinetics of MLS101: apparent terminal elimination half-life (t½) | Day 1 to Day 3 post-dose and end of study visit (Day 8)
Pharmacokinetics of MLS101: apparent total systemic clearance after oral administration (CL/F) | Day 1 to Day 3 post-dose and end of study visit (Day 8)
Pharmacokinetics of MLS101: apparent volume of distribution during the terminal phase (Vz/F) | Day 1 to Day 3 post-dose and end of study visit (Day 8)
Sensorial effects of MLS101 | Day 1 post-dose and end of study visit (Day 8)
  Using validated questionnaires, the nominal sensorial threshold dose of MLS101 will be identified. The nominal sensorial threshold dose is defined as the highest dose studied that is absent of clinically significant sensorial effects, and which would not interfere with the participant's ability to carry on with routine activities of daily living. Higher scores indicate presence of sensorial effects.
Cognitive function | Pre-dose (Day -1), Day 1 post-dose and end of study visit (Day 8)
  Using validated questionnaires and tools, cognitive function will be assessed and scores will be summarized for each visit, including observed values and change from baseline to evaluate the effects of MLS101 on participants' cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, Principal Investigator — Principal Investigator at CMAX Clinical Research Pty Ltd
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No